CLINICAL TRIAL: NCT06058234
Title: Prospective Study on Anti-Amyloid-β Monoclonal Antibodies Directed Against Amyloid for the Treatment of Alzheimer's Disease Coverage of Evidence Development (The Anti-Aβ mAb CED Study)
Brief Title: Medicare Anti-Aβ mAb Coverage With Evidence Development (CED) Study
Status: Recruiting | Type: Observational
Sponsor: Centers for Medicare and Medicaid Services/ Coverage and Analysis Group (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 99999999
Record Dates: First submitted 2023-09-08; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Mild Alzheimer's Disease; Mild Cognitive Impairment (MCI) Due to Alzheimer's Disease
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Monoclonal Antibodies Directed Against Amyloid for the Treatment of Alzheimer's Disease — FDA approved monoclonal antibodies directed against amyloid for the treatment of AD

SUMMARY:
The Anti-Aβ mAb CED Study is a prospective, longitudinal coverage with evidence development (CED) study using clinical data, patient assessments, and administrative claims data of the Medicare population, conducted in accordance to the National Coverage Determination (NCD) on Monoclonal Antibodies Directed Against Amyloid for the Treatment of Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
The Anti-Aβ mAb CED Study is conducted in accordance with the coverage criteria specified in the NCD for patients who have a clinical diagnosis of mild cognitive impairment (MCI) due to AD or mild AD dementia. The complete NCD decision memorandum is available on our website (https://www.cms.gov/medicare-coverage-database/view/ncacal-decisionmemo.aspx?proposed=N&ncaid=305).

Study Overview:

1. Clinicians will conduct a neurocognitive evaluation to determine patient eligibility by confirming a clinical diagnosis of MCI due to AD or mild AD dementia, and the presence of amyloid using biomarker testing including imaging (amyloid PET), cerebral spinal fluid (CSF) studies, and/or blood tests.
2. For all Medicare beneficiaries receiving anti-Aβ mAb treatment for MCI due to AD or mild AD dementia, the prescribing clinician will assess the patient's baseline clinical status by cognition and function assessments using validated tools appropriate for use in the MCI with AD and mild AD dementia populations and submit these data to the registry via the dedicated CMS CED submission portal every six months for up to 24 months (five total assessments).
3. In addition to performing the required cognition and function assessments, prescribing clinicians will need to report on the patient's use of anti-platelet and/or anti-coagulation therapy and whether the patient has developed new amyloid related imaging abnormalities (ARIA) since the last assessment data submission.

ELIGIBILITY:
Inclusion Criteria:

* Medicare patients with a clinical diagnosis of mild cognitive impairment due to Alzheimer's disease (AD) or mild AD dementia, both with confirmed presence of amyloid beta pathology consistent with AD.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medicare patients with a clinical diagnosis of mild cognitive impairment due to Alzheimer's disease (AD) or mild AD dementia, both with confirmed presence of amyloid beta pathology consistent with AD.
Sampling Method: Probability Sample
Enrollment: 8680 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in cognition | 24 months
  Cognition measured by the Montreal Cognitive Assessment (MoCA©) (score ranges from 0 to 30; higher scores are generally better).
Change in cognition | 24 months
  Cognition as measured by global Clinical Dementia Rating (CDR) (each of six domains ranges from 0 to 3; lower scores are generally better).
Change in function | 24 months
  Function as measured by global Clinical Dementia Rating (CDR) (each of six domains ranges from 0 to 3; lower scores are generally better).
Change in function | 24 months
  Function as measured by the Functional Activities Questionnaire (FAQ) (scores range from 0 to 30; lower scores are generally better).
Adverse Events (Harms) | 24 months
  Incidence of adverse events such as amyloid related imaging abnormalities (ARIA), stroke, infections.

CONTACTS AND LOCATIONS:
Locations (1):
- Centers for Medicare and Medicaid Services, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: medicare National Coverage Determination — https://www.cms.gov/medicare-coverage-database/view/ncacal-decision-memo.aspx?proposed=N&ncaid=305
- See also: Monoclonal Antibodies Directed Against Amyloid for the Treatment of Alzheimer's Disease CED Study Registry — https://qualitynet.cms.gov/alzheimers-ced-registry
- See also: Study Description — https://www.cms.gov/files/document/ced-study-description.pdf